CLINICAL TRIAL: NCT06765928
Title: A Multicenter, Single-arm Study of the Efficacy and Safety of Selinexor Combined With Venetoclax as Maintenance Therapy After Allogeneic Hematopoietic Stem Cell Transplantation for Acute Myeloid Leukemia/Myelodysplastic Syndrome
Brief Title: Selinexor Combined With Venetoclax Maintenance Therapy After Allo-HSCT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hu Xiaoxia, Principal Investigator, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJBMT-010
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: MDS; AML, Adult
Keywords: MDS/AML; allogeneic hematopoietic stem cell transplantation; maintenance therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — selinexor; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): Post allo-HSCT maintenance with selinexor in combination with venetoclax for intermediate to high-risk MDS/AML
  Interventions: Drug: selinexor in combination with venetoclax

INTERVENTIONS:
Drug: selinexor in combination with venetoclax — After allo-HSCT, intermediate-high risk MDS/AML patients are maintenanced with selinexor given in combination with venetoclax for 2 years
  Other Names: XPO1 inhibitor combined with Bcl-2 inhibitor

SUMMARY:
A multicenter, single-arm clinical study of evaluate the efficacy and safety of selinexor combined with venetoclax as maintenance therapy following allogeneic hematopoietic stem cell transplantation for acute myeloid leukemia patients.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is a curative treatment for intermediate- to high-risk acute myeloid leukemia (AML) and myelodysplastic syndromes (MDS).However, there are still some patients who relapse after transplantation, resulting in treatment failure. Therefore, post-transplantation maintenance therapy is needed for AML/MDS patients with poor prognosis to further reduce recurrence and prolong survival. In in vitro studies, XPO1 inhibitor combined with venetoclax was found to have a promising anti-leukemic effect, and venetoclax increased ROS levels in the bone marrow microenvironment and improved the post-transplant immune microenvironment. Accordingly, we propose to carry out XPO1 inhibitor combined with venetoclax as maintenance therapy after allo-HSCT in patients with intermediate- to high-risk AML/MDS.

There is a lack of prospective, controlled studies to clarify the efficacy and safety of XPO1 inhibitor combined with venetoclax as maintenance therapy after allo-HSCTin patients with intermediate- to high-risk AML/MDS, especially those with out specific gene mutation which would be targeted with commerically available inhibitors. Therefore, this multicenter, single-arm study is designed to assess the efficacy and safety of selinexor combined with venetoclax as maintenance therapy after intermediate to high-risk MDS/AML after allo-HSCT, with the aim of providing a reference for clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* de novo AML in the ELN2022 high-risk group or MDS in the IPSS-M intermediate-high/high/very-high risk group
* Age 18-75 years old, gender is not limited
* First hematopoietic stem cell transplant with at least one eligible donor
* ECOG physical status score of 0-2
* The subject has received an allogeneic hematopoietic stem cell transplant within 90-120 days and STR-PCR shows complete donor chimerism;
* Have appropriate organ function, and laboratory results within 7 days prior to the start of trial treatment need to meet the following criteria:

AST and ALT) ≤ 3x ULN; Total serum bilirubin ≤ 1.5x ULN unless the patient has Gilbert syndrome; patients with Gilbert-Meulengracht syndrome with bilirubin ≤ 3.0 times the upper limit of normal and direct bilirubin ≤ 1.5 times the upper limit of normal may be included; HB ≥ 70 g/L (had not received a red blood cell transfusion within 1 week prior to administration); ANC ≥ 0.8 x 10^9/L (had not received long-acting colony-stimulating factor (LACSF) within 1 week prior to administration and short-acting colony-stimulating factor (SACSF) within 3 days prior to administration); Platelet count ≥ 20 x 10^9/L (had not received a platelet transfusion within 1 week prior to administration); serum creatinine ≤ 1.5x ULN or creatinine clearance ≥ 60 mL/min; Coagulation function: International Normalized Ratio (INR) ≤1.5×ULN, Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN; Left ventricular ejection fraction (LVEF) ≥45%;

* Life expectancy ≥ 12 weeks;
* Voluntarily sign the informed consent form and understand and comply with the requirements of the study.

Exclusion Criteria:

* bone marrow examination after allo-HSCT suggestive of relapse or measurable residual disease (MRD) before the initiation of maintenance therapy;
* Other malignant tumors within 5 years prior to screening, except adequately treated carcinoma in situ of the cervix, basal cell or squamous epithelial cell skin cancers, post-radical thyroid cancer, and post-radical ductal carcinoma in situ;
* Current active cardiovascular disease of clinical significance, such as uncontrolled arrhythmias, uncontrolled hypertension, congestive heart failure, any grade 3 or 4 heart disease as determined by the New York Heart Association (NYHA) functional class, or a history of myocardial infarction within the 6 months prior to screening;
* Other serious medical conditions that may limit the patient's participation in this trial (e.g., active infection, uncontrolled diabetes);
* Known HIV infection, or chronic infection with hepatitis B virus (HBsAg-positive) or hepatitis C virus (anti-HCV-positive) that cannot be controlled by medications;
* Patients with other tumors in combination, not cured;
* Patients with neurologic or psychiatric disorders; clinically significant active cerebrovascular disease (e.g., cerebral edema, posterior reversible encephalopathy syndrome);
* Those who are allergic to the test drug;
* Those who are unable to understand or comply with the study protocol or are unable to sign the informed consent form;
* Those who have received other maintenance drugs after hematopoietic stem cell transplantation or have the desire to receive other maintenance therapy;
* Participation in other clinical studies within 3 months prior to screening that have not interfered with the safety and efficacy of the study drug as assessed by the investigator is permitted for inclusion in the study, e.g., non-interventional observational studies;
* Patients who, in the investigator's judgment and/or clinical criteria, have contraindications to any of the study procedures or have other medical conditions that may place them at unacceptable risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival | through study completion, an average of 2 year
  disease progression or death as a result of any causes

SECONDARY OUTCOMES:
Overall survival | through study completion, an average of 2 year
  death as a result of any causes
Non-relapse survial | through study completion, an average of 2 year
  death without disease progression or relapse

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital of Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China